CLINICAL TRIAL: NCT03315936
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses of BI 894416 in Healthy Male Subjects (Single-blind, Partially Randomised, Placebo-controlled Parallel Group Design)
Brief Title: This Study in Healthy Men Tests How Different Doses of BI 894416 Are Taken up in the Body and How Well BI 894416 is Tolerated
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1371-0001; 2016-003470-40 (EudraCT Number)
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Placebo matching BI 894416 (SRD Part) (Placebo Comparator): Single Rising Dose (SRD) Part
  Interventions: Drug: Placebo
- BI 894416 3 milligram (mg) (Experimental): SRD Part
  Interventions: Drug: BI 894416
- BI 894416 10 mg (Experimental): SRD Part
  Interventions: Drug: BI 894416
- BI 894416 20 mg (Experimental): SRD Part
  Interventions: Drug: BI 894416
- BI 894416 30 mg (Experimental): SRD Part
  Interventions: Drug: BI 894416
- BI 894416 40 mg (Experimental): SRD Part
  Interventions: Drug: BI 894416
- BI 894416 54 mg (Experimental): SRD Part
  Interventions: Drug: BI 894416
- BI 894416 70 mg (Experimental): SRD Part
  Interventions: Drug: BI 894416
- BI 894416 10mg tb / 10mg PfOS / 40mg tb (Experimental): BI 894416 10 mg tablet (tb) / BI 894416 10 mg powder for oral solution (PfOS) / BI 894416 4*10 mg tablets.
  Relative bioavailability (rel BA) part
  Interventions: Drug: BI 894416
- BI 894416 10mg PfOS / 10mg tb / 40mg tb (Experimental): BI 894416 10 mg powder for oral solution (PfOS) / BI 894416 10 mg tablet (tb) / BI 894416 4*10 mg tablets.
  Relative bioavailability (rel BA) part.
  Interventions: Drug: BI 894416

INTERVENTIONS:
Drug: BI 894416 — powder for oral solution
  Arms: BI 894416 10 mg; BI 894416 10mg PfOS / 10mg tb / 40mg tb; BI 894416 10mg tb / 10mg PfOS / 40mg tb; BI 894416 20 mg; BI 894416 3 milligram (mg); BI 894416 30 mg; BI 894416 40 mg; BI 894416 54 mg; BI 894416 70 mg
Drug: Placebo — Oral solution
  Arms: Placebo matching BI 894416 (SRD Part)
Drug: BI 894416 — Tablet
  Arms: BI 894416 10mg PfOS / 10mg tb / 40mg tb; BI 894416 10mg tb / 10mg PfOS / 40mg tb

SUMMARY:
This first-in man trial is designed to investigate the safety and tolerability of BI 894416 in healthy male subjects following oral administration of single rising doses.

Pharmacokinetics (PK) including dose proportionality after single dosing of BI 894416 as oral solution will be explored, the investigation of PK of BI 894416 as tablet formulation and the exploration of relative bioavailability of BI 894416 as tablet formulation compared to oral solution.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)),12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 45 years (incl.)
* Body Mass Index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG) and including the neurological examination) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

In addition, the following trial-specific exclusion criteria apply:

* History of relevant neurological disorder affecting the peripheral or central nervous system (this includes, but is not limited to: stroke, epilepsy, inflammatory or atrophic diseases affecting the nervous system, cluster headache or any cancer of the nervous system)
* History of immunological disease except allergy not relevant to the trial (such as mild hay fever or dust mite allergy) and except asthma in childhood or adolescence
* History of cancer (other than successfully treated basal cell carcinoma)
* Within 10 days prior to administration of trial medication, use of any drug that could reasonably inhibit platelet aggregation or coagulation (e.g., acetylsalicylic acid)
* Male subjects with woman of child bearing potential (WOCBP) partner who are unwilling to use male contraception (condom or sexual abstinence) from time point of administration of trial medication until 30 days thereafter.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single rising dose (SRD) part was designed as single-blind, partially randomized within dose groups, placebo-controlled, parallel-group design and relative bioavailability (rel BA) part was an open-label, randomized two-way crossover followed by a fixed sequence design in healthy volunteers.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants attended specialized site which would ensure that all participants met all inclusion/exclusion criteria. Participants were not to be entered/randomised to trial treatment if any one of the specific entry criteria were not met.
Groups:
- Placebo Matching BI 894416 (SRD Part): Participants were orally administered single dose of placebo solution matching to BI 894416 with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) in SRD Part.
- BI 894416 3 Milligram (mg) (SRD Part): Participants were administered single dose of BI 894416 3 milligram (mg) powder for oral solution (PfOS) with 240 mL of water after an overnight fast of at least 10 hours (h) in SRD Part.
- BI 894416 10 mg (SRD Part): Participants were administered single dose of BI 894416 10 mg powder for oral solution with 240 mL of water after an overnight fast of at least 10 h in SRD Part.
- BI 894416 20 mg (SRD Part): Participants were administered single dose of BI 894416 20 mg powder for oral solution with 240 mL of water after an overnight fast of at least 10 h in SRD Part.
- BI 894416 30 mg (SRD Part): Participants were administered single dose of BI 894416 30 mg powder for oral solution with 240 mL of water after an overnight fast of at least 10 h in SRD Part.
- BI 894416 40 mg (SRD Part): Participants were administered single dose of BI 894416 40 mg powder for oral solution with 240 mL of water after an overnight fast of at least 10 h in SRD Part.
- BI 894416 54 mg (SRD Part): Participants were administered single dose of BI 894416 54 mg powder for oral solution with 240 mL of water after an overnight fast of at least 10 h in SRD Part.
- BI 894416 70 mg (SRD Part): Participants were administered single dose of BI 894416 70 mg powder for oral solution with 240 mL of water after an overnight fast of at least 10 h in SRD Part.
- BI 894416 10mg tb / 10mg PfOS / 40mg tb: Participants were administered single dose of BI 894416 10 mg tablet (tb) in period 1 followed by BI 894416 10 mg powder for oral solution in period 2 followed by BI 894416 4*10 mg tablets in period 3. Dosages for all periods were administered with 240 mL of water after an overnight fast of at least 10 h. Treatments in period 1 and 2 were separated by a wash-out period of at least 6 days and treatments in periods 2 and 3 were separated by a wash-out period of at least 10 days, in rel BA Part.
- BI 894416 10mg PfOS / 10mg tb / 40mg tb: Participants were administered single dose of BI 894416 10 mg powder for oral solution in period 1 followed by BI 894416 10 mg tablet (tb) in period 2 followed by BI 894416 4*10 mg tablets in period 3. Dosages for all periods were administered with 240 mL of water after an overnight fast of at least 10 h. Treatments in period 1 and 2 were separated by a wash-out period of at least 6 days and treatments in periods 2 and 3 were separated by a wash-out period of at least 10 days, in rel BA Part.
Period: Period 1
Arm/Group | Placebo Matching BI 894416 (SRD Part) | BI 894416 3 Milligram (mg) (SRD Part) | BI 894416 10 mg (SRD Part) | BI 894416 20 mg (SRD Part) | BI 894416 30 mg (SRD Part) | BI 894416 40 mg (SRD Part) | BI 894416 54 mg (SRD Part) | BI 894416 70 mg (SRD Part) | BI 894416 10mg tb / 10mg PfOS / 40mg tb | BI 894416 10mg PfOS / 10mg tb / 40mg tb
Started (Started are treated) | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Placebo Matching BI 894416 (SRD Part) | BI 894416 3 Milligram (mg) (SRD Part) | BI 894416 10 mg (SRD Part) | BI 894416 20 mg (SRD Part) | BI 894416 30 mg (SRD Part) | BI 894416 40 mg (SRD Part) | BI 894416 54 mg (SRD Part) | BI 894416 70 mg (SRD Part) | BI 894416 10mg tb / 10mg PfOS / 40mg tb | BI 894416 10mg PfOS / 10mg tb / 40mg tb
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Placebo Matching BI 894416 (SRD Part) | BI 894416 3 Milligram (mg) (SRD Part) | BI 894416 10 mg (SRD Part) | BI 894416 20 mg (SRD Part) | BI 894416 30 mg (SRD Part) | BI 894416 40 mg (SRD Part) | BI 894416 54 mg (SRD Part) | BI 894416 70 mg (SRD Part) | BI 894416 10mg tb / 10mg PfOS / 40mg tb | BI 894416 10mg PfOS / 10mg tb / 40mg tb
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This subject set included all subjects who received at least 1 dose of BI 894416 or placebo.
Groups:
- Placebo Matching BI 894416 (SRD Part): Participants were orally administered single dose of placebo solution matching to BI 894416 with 240 mL of water after an overnight fast of at least 10 hours (h) in SRD Part.
- Total: Total of all reporting groups
Arm/Group | Placebo Matching BI 894416 (SRD Part) | BI 894416 3 Milligram (mg) (SRD Part) | BI 894416 10 mg (SRD Part) | BI 894416 20 mg (SRD Part) | BI 894416 30 mg (SRD Part) | BI 894416 40 mg (SRD Part) | BI 894416 54 mg (SRD Part) | BI 894416 70 mg (SRD Part) | BI 894416 10mg tb / 10mg PfOS / 40mg tb | BI 894416 10mg PfOS / 10mg tb / 40mg tb | Total
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 68
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.8 (7.3) | 33.2 (7.3) | 33.5 (6.4) | 35.7 (7.1) | 33.7 (7.0) | 38.2 (6.3) | 34.3 (5.5) | 34.2 (9.1) | 31.7 (8.3) | 30.5 (6.9) | 33.9 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 13 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 66
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 14 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 67
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Drug-related Adverse Events in SRD Part
Description: Percentage of participants with drug-related adverse events (AEs) in SRD part. Percentages are calculated using total number of subjects per treatment as the denominator. Percentages were rounded up to 1 decimal places.
Time Frame: From drug administration until end of the trial, up to 17 days.
Population: Treated set (TS): This subject set included all subjects who received at least 1 dose of BI 894416 or placebo.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Matching BI 894416 (SRD Part) | BI 894416 3 Milligram (mg) (SRD Part) | BI 894416 10 mg (SRD Part) | BI 894416 20 mg (SRD Part) | BI 894416 30 mg (SRD Part) | BI 894416 40 mg (SRD Part) | BI 894416 54 mg (SRD Part) | BI 894416 70 mg (SRD Part)
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Percentage of participants | 0.0 | 0.0 | 0.0 | 33.3 | 16.7 | 0.0 | 16.7 | 16.7

2. Secondary Outcome: Area Under the Concentration-time Curve of BI 894416 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-inf) in SRD Part
Description: Area under the concentration-time curve of BI 894416 in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf) in SRD part is presented.
Time Frame: Pharmacokinetic samples were collected at 2 hours (h) prior drug administration and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 34, 48, 72, 96, 168 h after drug administration.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): This subject set included all subjects of the treated set who provided at least 1 PK parameter that was not excluded because of an important protocol deviation relevant to the statistical evaluation of PK endpoints or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole (nmol) * hour (h) / Litre (L)
Arm/Group | BI 894416 3 Milligram (mg) (SRD Part) | BI 894416 10 mg (SRD Part) | BI 894416 20 mg (SRD Part) | BI 894416 30 mg (SRD Part) | BI 894416 40 mg (SRD Part) | BI 894416 54 mg (SRD Part) | BI 894416 70 mg (SRD Part)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
nanomole (nmol) * hour (h) / Litre (L) | 345 (34.9) | 640 (101.0) | 1470 (96.7) | 3270 (27.1) | 6020 (20.6) | 7210 (28.1) | 11400 (29.6)

3. Secondary Outcome: Maximum Measured Concentration of BI 894416 in Plasma (Cmax) in SRD Part
Description: Maximum measured concentration of BI 894416 in plasma (Cmax) in SRD part is presented.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole (nmol)/Litre (L)
Arm/Group | BI 894416 3 Milligram (mg) (SRD Part) | BI 894416 10 mg (SRD Part) | BI 894416 20 mg (SRD Part) | BI 894416 30 mg (SRD Part) | BI 894416 40 mg (SRD Part) | BI 894416 54 mg (SRD Part) | BI 894416 70 mg (SRD Part)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
nanomole (nmol)/Litre (L) | 55.4 (11.1) | 161.0 (37.5) | 352.0 (26.9) | 527.0 (31.3) | 1170.0 (26.4) | 1240.0 (23.0) | 2130.0 (16.7)

4. Secondary Outcome: Area Under the Concentration-time Curve of BI 894416 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz) in Rel BA Part
Description: Area under the concentration-time curve of BI 894416 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) in rel BA part is presented. "BI 894416 40 mg tb" arm was compared in a descriptive fashion with other dose groups without statistical analysis.
Time Frame: Pharmacokinetic samples were collected at 2 hours (h) prior drug administration and at 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 h after drug administration.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole (nmol) * hour (h)/Litre (L)
Groups:
- BI 894416 10 mg tb (T): Participants were administered single dose of BI 894416 10 mg tablet with 240 mL of water after an overnight fast of at least 10 h in rel BA part.
- BI 894416 10 mg PfOS (R): Participants were administered single dose of BI 894416 10 mg powder for oral solution with 240 mL of water after an overnight fast of at least 10 h in rel BA part.
- BI 894416 40 mg tb: Participants were administered single dose of BI 894416 4*10 mg tablets with 240 mL of water after an overnight fast of at least 10 h in rel BA part.
Arm/Group | BI 894416 10 mg tb (T) | BI 894416 10 mg PfOS (R) | BI 894416 40 mg tb
Number analyzed (Participants) | 12 | 12 | 12
nanomole (nmol) * hour (h)/Litre (L) | 941 (95.2) | 853 (89.0) | 5870 (61.2)
Statistical Analysis 1: Comparison: BI 894416 10 mg tb (T) vs BI 894416 10 mg PfOS (R); The analysis of variance (ANOVA) model on the logarithmic scale including 'sequence', 'period', and 'treatment' as fixed effects and 'subject within sequence' as random effect. No hypothesis was tested and no acceptance range was specified. This was an intra-individual assessment and actually 12 subjects were analyzed; Test type: Other; geometric mean (gMean) ratio (T/R) % = 110.31, 90% CI 2-sided [100.73 to 120.79] — To get, gMean ratio (T/R) and confidence interval, least square estimates of log-transformed PK endpoint for T and R were back transformed to original scale. Intra-individual geometric coefficient of variation (%) = 12.3

5. Secondary Outcome: Area Under the Concentration-time Curve of BI 894416 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-inf) in Rel BA Part
Description: Area under the concentration-time curve of BI 894416 in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf) in rel BA part is presented. "BI 894416 40 mg tb" arm was compared in a descriptive fashion with other dose groups without statistical analysis.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole (nmol) * hour (h)/Litre (L)
Arm/Group | BI 894416 10 mg tb (T) | BI 894416 10 mg PfOS (R) | BI 894416 40 mg tb
Number analyzed (Participants) | 12 | 12 | 12
nanomole (nmol) * hour (h)/Litre (L) | 975 (97.5) | 879 (90.4) | 6060 (63.5)
Statistical Analysis 1: Comparison: BI 894416 10 mg tb (T) vs BI 894416 10 mg PfOS (R); The analysis of variance (ANOVA) model on the logarithmic scale including 'sequence', 'period', and 'treatment' as fixed effects and 'subject within sequence' as random effect. No hypothesis was tested and no acceptance range was specified. This was an intra-individual assessment and actually only 12 subjects were analyzed; Test type: Other; gMean ratio (T/R) % = 110.83, 90% CI 2-sided [101.20 to 121.38] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Maximum Measured Concentration of BI 894416 in Plasma (Cmax) in Rel BA Part
Description: Maximum measured concentration of BI 894416 in plasma (Cmax) in rel BA part is presented. "BI 894416 40 mg tb" arm was compared in a descriptive fashion with other dose groups without statistical analysis.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole (nmol)/Litre (L)
Arm/Group | BI 894416 10 mg tb (T) | BI 894416 10 mg PfOS (R) | BI 894416 40 mg tb
Number analyzed (Participants) | 12 | 12 | 12
nanomole (nmol)/Litre (L) | 199 (39.5) | 180 (53.4) | 1160 (39.2)
Statistical Analysis 1: Comparison: BI 894416 10 mg tb (T) vs BI 894416 10 mg PfOS (R); [analysis description as in outcome 5, analysis 1]; Test type: Other; gMean ratio (T/R) % = 110.46, 90% CI 2-sided [89.74 to 135.96] — To get, gMean ratio (T/R) and confidence interval, least square estimates of log-transformed PK endpoint for T and R were back transformed to original scale. Intra-individual geometric coefficient of variation (%) = 28.6

ADVERSE EVENTS:
Time Frame: For SRD part: From drug administration until end of the trial, up to 17 days. For rel BA part: From drug administration until end of the trial, up to 54 days.
Description: Treated set (TS): This subject set included all subjects who received at least 1 dose of BI 894416 or placebo.
Arm/Group | Placebo Matching BI 894416 (SRD Part) | BI 894416 3 Milligram (mg) (SRD Part) | BI 894416 10 mg (SRD Part) | BI 894416 20 mg (SRD Part) | BI 894416 30 mg (SRD Part) | BI 894416 40 mg (SRD Part) | BI 894416 54 mg (SRD Part) | BI 894416 70 mg (SRD Part) | BI 894416 10 mg PfOS (R) | BI 894416 10 mg tb (T) | BI 894416 40 mg tb
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/14 | 2/6 | 2/6 | 5/6 | 2/6 | 2/6 | 1/6 | 2/6 | 4/12 | 3/12 | 4/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matching BI 894416 (SRD Part) (N=14) | BI 894416 3 Milligram (mg) (SRD Part) (N=6) | BI 894416 10 mg (SRD Part) (N=6) | BI 894416 20 mg (SRD Part) (N=6) | BI 894416 30 mg (SRD Part) (N=6) | BI 894416 40 mg (SRD Part) (N=6) | BI 894416 54 mg (SRD Part) (N=6) | BI 894416 70 mg (SRD Part) (N=6) | BI 894416 10 mg PfOS (R) (N=12) | BI 894416 10 mg tb (T) (N=12) | BI 894416 40 mg tb (N=12)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral mucosal eruption (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral papule (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 1 | 2 | 0 | 1 | 1 | 2 | 2 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Ocular discomfort (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/36/NCT03315936/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/36/NCT03315936/SAP_001.pdf